CLINICAL TRIAL: NCT00558935
Title: The Effect of Alcohol on ABCA1 Expression and Lipid Metabolism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was found that 20g of alcohol daily had no effect on ABCA1 expression or HDL levels.
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 24/06
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Type 2 Diabetes; Heart Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Dietary Supplement: Red Wine — 20g alcohol daily/red wine for 4 weeks

SUMMARY:
The purpose of this study is to investigate the effects of red wine on ABCA1 levels

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Aged 18-65 years
* Free of overt coronary disease
* BMI < 35
* Fasting plasma glucose <6.1 mmol
* Unmedicated
* No major illness

Exclusion Criteria:

* Unable to give informed consent
* Smokers
* Participants with alcoholism

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
measurements of dyslipidemia | 2 years

SECONDARY OUTCOMES:
lipid functionality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn A Kingwell, PhD, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Baker Heart Research Institute, Melbourne, Victoria, Australia